CLINICAL TRIAL: NCT07009899
Title: BCMA Bispecific Antibody Therapy for Post-BCMA CAR T-Cell Therapy Relapse (RECLAIM)
Acronym: RECLAIM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Dhakal, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00056695
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Bispecific Antibody; BCMA; BCMA CAR T-Cell Therapy; linvoseltamab; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Linvoseltamab Administration (Experimental): Linvoseltamab intravenous (IV) will be initially administered to all patients as a step-up dosing regimen during the first two weeks of Cycle 1 (Weeks 1 and 2; 5 mg on Cycle 1 Day 1 and 25 mg on Cycle 1 Day 8) in an inpatient setting. Starting with Cycle 1 Day 15 (Week 3), linvoseltamab 200 mg will be administered once a week until the end of Cycle 3 (Week 12) followed by once every two weeks (Days 1 and 15) during Cycles 4 through 6 (Weeks 13 through 24). From Cycle 7 Day 1 (Week 25) until disease progression, linvoseltamab 200 mg will be administered once every four weeks.
  Interventions: Drug: Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — Linvoseltamab is a human IgG4-based bsAb that binds to CD3, a T-cell antigen associated with the TCR complex, and BCMA, which is expressed on the surface of malignant MM B-lineage cells, as well as late-stage B cells and plasma cells.

SUMMARY:
This is a single-center, single-arm, phase 2 study designed to evaluate the efficacy and safety of linvoseltamab in multiple myeloma (MM) patients who relapsed following BCMA CAR T-cell therapy, whether standard of care or investigational.

DETAILED DESCRIPTION:
This is a single-center, single-arm, phase 2 study designed to evaluate the efficacy and safety of linvoseltamab in multiple myeloma (MM) patients who relapsed following BCMA CAR T-cell therapy, whether standard of care or investigational. The primary objective is to assess overall response rate (ORR) in patients treated with linvoseltamab.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status criteria of 0-3.
3. Received any standard of care or investigational BCMA CAR T-cell therapy as their last line of therapy ≥ 6 months prior to enrollment.

   a. Note: Up to 15% of patients who are < 6 months out from their standard of care of investigational BCMA CAR T-cell therapy will be included in the study as long as i) their bone marrow biopsy sample tests positive for BCMA expression by immunohistochemistry and ii) they have stem cells available for a stem cell boost therapy prior to linvoseltamab administration.
4. Must have measurable disease for response assessment as per the IMWG response assessment criteria.

   a. Note: if a patient does not have measurable serum M or free light chain, evidence of measurable disease by imaging is acceptable (e.g., extramedullary disease, new lesions).
5. Adequate hepatic function as defined below:

   1. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
6. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Previously on a BCMA-directed therapy other than BCMA CAR T-cell therapy (e.g., BCMA bispecific antibody, BCMA antibody drug conjugate) or T cell engaging therapy (e.g., GPRC5D bispecific antibody, GPRC5D CAR T-cell therapy).
2. History of neurodegenerative condition, Central Nervous System (CNS) movement disorder, or patients with a history of seizure within 12 months prior to study enrollment.
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
4. Prior organ transplant requiring immunosuppressive therapy.
5. Known to be human immunodeficiency virus (HIV) positive.
6. Known to have hepatitis A, B, or C active infection.
7. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
8. Concurrent hematologic or non-hematologic malignancy requiring treatment (other than multiple myeloma and secondary amyloidosis).
9. Cardiac syncope, uncompensated New York Heart Association (NYHA) Class 3 or 4 congestive heart failure, myocardial infarction within the previous six months, unstable angina pectoris, clinically significant repetitive ventricular arrhythmias despite antiarrhythmic treatment, cardiac ejection fraction < 40% by echocardiogram or multi-gated acquisition (MUGA) scan, severe orthostatic hypotension, or clinically important autonomic disease.
10. Major surgery within 14 days prior to start of study treatment (Note: vertebroplasty and kyphoplasty are not considered major surgery).
11. Infection requiring systemic antibiotic therapy or other serious infection within 14 days prior to start of study treatment.
12. Active treatment in other clinical trials, including those where a subject received an investigational drug within 30 days or five half-lives of the investigational drug prior to start of study treatment, whichever is longer.
13. Any clinically significant, uncontrolled medical conditions that, in the investigator's opinion, would expose the subject to excessive risk or may interfere with compliance or interpretation of the study results.
14. Pregnant or breastfeeding women.
15. Women of childbearing potential (WOCBP) or sexually active men who are unwilling to practice highly effective contraception prior to the start of study therapy, during the study, and for at least 6 months after the last dose of the study drug.

    1. WOCBP are defined as women who are fertile following menarche until becoming postmenopausal (defined as no menses for 12 months without an alternative medical cause), unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
    2. Male study participants with WOCBP partners are required to use condoms unless they are vasectomized or practice sexual abstinence. Male study participants should not donate sperm during the study, and for at least 6 months after the last dose
16. Highly effective contraceptive measures include stable use of combined (estrogen and progestogen-containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated two or more menstrual cycles prior to screening; intrauterine device; intrauterine hormone-releasing system; bilateral tubal ligation; vasectomized partner (provided that the vasectomized partner is the sole sexual partner of the WOCBP study participant); and or sexual abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 15 months
  This is the number of subjects who have a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Meera Mohan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No